CLINICAL TRIAL: NCT05961111
Title: An Open, Single-armed, Clinical Safety and Efficacy Study on Oncolytic Virus Injection (R130 OV) for the Treatment of Advanced Solid Tumors
Brief Title: A Clinical Study on Oncolytic Virus Injection (R130 OV) for the Treatment of Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Yunying Medical Technology (Industry)
Collaborators: Linyi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYCH-R130
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sarcoma; Carcinoma; Digestive Cancer; Breast Cancer; Lung Cancer; Brain Cancer; Melanoma; Gynecologic Cancer; Head and Neck Cancer; Kidney Cancer
Keywords: Oncolytic virus; Herpes simplex virus type 1
MeSH Terms: conditions — Sarcoma; Carcinoma; Gastrointestinal Neoplasms; Breast Neoplasms; Lung Neoplasms; Brain Neoplasms; Melanoma; Head and Neck Neoplasms; Kidney Neoplasms | interventions — Oncolytic Virotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R130 Treatment Group (Experimental): Every 7-14 days,1-2 ml R130 （concentration of 1x10^8 plaque-forming Units/mL,PFU/mL）will be injected intratumoral or intraperitoneal in patients with advanced solid tumors
  Interventions: Drug: Recombinant oncolytic herpes simplex virus type 1 (R130)

INTERVENTIONS:
Drug: Recombinant oncolytic herpes simplex virus type 1 (R130) — R130, a modified herpes simplex virus-Ⅰ (HSV-1) containing the gene coding for anti-CD3 scFv/CD86/PD1/HSV2-US11
  Other Names: Oncolytic virus

SUMMARY:
20 participants are expected to be enrolled for this open，Single-armed clinical trial to evaluate the safety and efficacy of the recombinant herpes simplex virus Ⅰ, R130 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid tumors clearly diagnosed by histology and/or cytology.
2. Failure of standard treatment or patient unwillingness to receive other antitumor therapy.
3. Age 18 to 75 years.
4. Subjects with ECoG score of 0-2.
5. Expected survival of 3 months or more.
6. Have at least one measurable lesion (according to RECIST 1.1 criteria) that is amenable to intratumoral or intraperitoneal drug delivery.
7. Subjects must have appropriate organ function, and laboratory tests during the screening period must meet the following requirements: a) absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets (PLT) ≥ 80 × 109/L, and hemoglobin (Hb) ≥ 85 g/L; b) serum creatinine (Cr) and blood urea nitrogen (BUN) within 1.5 times the upper limit of normal values; c) serum c) serum total bilirubin (TBIL) ≤ 2 times the upper limit of normal values; d) glutamic aminotransferase (ALT) and glutamic oxalacetic aminotransferase (AST) ≤ 2.5 times the upper limit of normal values; subjects with liver metastases do not exceed 5 times the upper limit of normal values; e) activated partial thromboplastin time (APTT), prothrombin time (PT) within 1.5 times the upper limit of normal values.
8. No absolute or relative centasis contraindiction.
9. Eligible patients of childbearing potential must agree to use a reliable method of contraception with their partner for the duration of the trial and for at least 180 days after the last dose; female patients of childbearing potential must have a negative urine pregnancy test within 7 days prior to enrollment.
10. Subjects voluntarily sign an informed consent form and are in good compliance.

Exclusion Criteria:

1. Have had any serious adverse reactions associated with immunotherapy.
2. Subjects with any severe and/or uncontrolled disease, including: a) poorly controlled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg); b) suffering from class I or higher myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470 ms and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification); c) active or uncontrolled severe infection (≥ CTCAE grade 2 infection); d) Patients with previous organ transplantation, bone marrow transplantation (hematopoietic stem cell transplantation) and severe immune deficiency; e) Urine routine suggesting urine protein ≥++ and confirmed 24-hour urine protein quantification > 1.0 g.
3. Patients with past history of type I diabetes mellitus or HIV.
4. Severe abnormalities in thyroid and cortisol testing; active, known or suspected autoimmune disease requiring systemic therapy.
5. Patients with severe prior interstitial lung changes (as determined by the investigator).
6. Patients with active tuberculosis and a strong positive OT test.
7. Patients with active bleeding or severe coagulation dysfunction.
8. Have had antitumor therapy, including endocrine, chemotherapy, radiotherapy, targeted therapy, immunotherapy and antitumor herbal therapy, 4 weeks prior to the first dose.
9. Have not recovered to CTCAE 4.0 grade rating 0 or 1 level of toxicity after previous antineoplastic therapy.
10. Current active hepatitis B, active hepatitis C, immunodeficiency virus or other active infection of clinical significance.
11. Patients who have undergone surgery of grade 3 or higher or whose surgical wounds have not healed within 4 weeks prior to enrollment.
12. Pregnant, lactating and planning to have children within six months.
13. Subjects who, in the judgment of the investigator, are unsuitable for participation in this trial for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Subject incidence of adverse events | Up to 6 months
  To characterize the safety profile of R130 injection in patients with advanced solid tumors as measured by the incidence of Grade ≥ 3 Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE v5.0),such as fever, fatigue, flu like symptoms, chills, Injection site reaction,etc.
Subject incidence of laboratory abnormalities | Up to 1 month
Systemic Immune Response | Up to 6 months
  Detection of increased systemic immune Response markers in sera (IL2,IL4,IL6,IL8,IL10,TNFa，IFNγ, etc.) and peripheral blood mononuclear cells by multi-Color fluorescence-activated cell sorting (FACS)

SECONDARY OUTCOMES:
Disease Assessment for Disease Control Rate | Every 10 weeks for 12 months
  CT will be performed to evaluate the efficacy endpoints of DCR by the investigator with RECIST v1.1 and iRECIST. DCR (proportion of patients) = with CR +PR +SD /CR + PR +SD + PD.
Disease Assessment for Duration of Response | Every 10 weeks for 12 months
  The time length between the first confirmed objective response per RECIST 1.1 to the treatment and the subsequent disease progression per RECIST 1.1
Quality of Life Assessment | Every 6 weeks for 12 months
  Comparison of patients' quality of life before and after R130 treatment as assessed by the EORTC QLQ-30 (V3.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Linyi Central Hospital, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided